CLINICAL TRIAL: NCT02716701
Title: Effects of Exercise on Brain Structure and Function in Multiple Sclerosis
Brief Title: Exercise in Multiple Sclerosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funding
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 4607-B
Record Dates: First submitted 2016-03-10; First posted 2016-03-23 (Estimated); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Multiple Sclerosis
Keywords: Exercise
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): Subjects will wear a wristband activity tracker to monitor their physical activity and will be asked to increase their activity level, with a goal of at least doubling their average daily activity (steps)
  Interventions: Behavioral: Exercise Group; Other: wristband activity tracker
- Control Group (Active Comparator): Subjects will wear a wristband activity tracker to monitor their physical activity and will not be encouraged to increase their activity level
  Interventions: Other: Control Group; Other: wristband activity tracker

INTERVENTIONS:
Behavioral: Exercise Group
  Arms: Exercise Group
Other: Control Group
  Arms: Control Group
Other: wristband activity tracker

SUMMARY:
Exercise therapy in MS patients has proven benefits on mobility, mood, motor function and quality of life. While the beneficial effects of exercise on cardiovascular and musculoskeletal function are well known, there has recently been increased focus on the positive effects of exercise on brain structure and function. The goal of this study is to determine whether exercise can promote beneficial changes in brain function in MS patients.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a chronic, disabling neurologic disease characterized by damage to myelin and axons in the central nervous system (CNS). Current therapy for MS primarily consists of immunomodulatory drugs aimed at preventing future CNS injury; no treatments are currently available to repair existing damage, and symptomatic treatments to improve neurological function are quite limited. Rehabilitation approaches, such as exercise, have long been a staple of MS therapy. Exercise therapy in MS patients has proven benefits on mobility, mood, motor function and quality of life. While the beneficial effects of exercise on cardiovascular and musculoskeletal function are well known, there has recently been increased focus on the positive effects of exercise on brain structure and function. The overall aim of this proposal is to determine whether exercise can promote beneficial changes in brain function in MS patients. The investigator's central hypothesis is that cardiovascular exercise alters both brain structure and brain function in MS patients, and that these changes can be identified and monitored via imaging techniques that evaluate regional brain volumes and functional connectivity. When brain activity measured at one area fluctuates in a coherent manner with that recorded in a different area, those brain regions are considered to be functionally connected. Using resting-state magnetoencephalography (MEG), the investigator's laboratory has demonstrated that these patterns of correlated brain activity are abnormal in MS patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with a confirmed diagnosis of MS by revised McDonald criteria
* Age ≥ 18 years
* Expanded Disability Status Scale (EDSS) 0-6.0, inclusive.
* Able to understand the consent process, and the use of the wristband activity tracker.
* Sedentary by self-report (answers no to the question: "Do you exercise regularly?"
* Willing to make sincere effort to comply with the study objective of increasing their physical activity as much as possible (with goal of at least 100% increase) and to maintain that increased activity level for six months (if randomized to the exercise group).

Exclusion Criteria:

* Current serious medical condition which would likely limit subject's ability to achieve sustained increase in physical activity, or put them at risk for doing so in the investigators' opinion (e.g. significant cardiovascular or respiratory disease, cancer, cancer, orthopedic disease, etc)
* Subjects that have a central nervous system disorder (in addition to MS) that is not considered secondary to MS
* Subjects that have implanted metal, pacemaker, etc. that may interfere with the MEG/MRI scan or who are otherwise unable to complete the MEG/MRI scan procedure without sedation (e.g. due to claustrophobia, obesity)
* weight > 300 pounds

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-01; Primary Completion 2020-08-12 (Actual); Study Completion 2020-08-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline in brain structure as measured by magnetic resonance imaging scans at 7 months | 7 months
  Magnetic resonance imaging (MRI) scans will be done at 1 month (baseline) and 7 months after subjects begin wearing a wristband activity tracker.
Change from baseline in brain structure as measured by magnetoencephalography (MEG) scans at 7 months | 7 months
  MEG scans will be done at 1 month (baseline) and 7 months after subjects begin wearing a wristband activity tracker

CONTACTS AND LOCATIONS:
Overall Officials: Adam F Carpenter, MD, Principal Investigator — Minneapolis Veterans Affairs Medical Center
Locations (1):
- VA Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No